CLINICAL TRIAL: NCT06454604
Title: Development of a Novel Virtual Reality Treatment for Emerging Adults With ADHD
Brief Title: Virtual Reality Treatment for Emerging Adults With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Joshua M. Langberg, Ph.D., Professor of Psychology, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2023001005; R61MH131632-01 (NIH)
Record Dates: First submitted 2024-05-31; First posted 2024-06-12 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Virtual reality
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Parallel group randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR Passthrough (Active Comparator): Participants in this condition wear the same VR headset as participants in the in the other arms. However, they see directly through to their laptop and are not emersed in the virtual world.
  Interventions: Behavioral: Meta Quest 3 VR Headset with noise cancelling headphones
- Virtual Reality (Experimental): Participants in this condition wear the virtual reality headset. They are emersed in a virtual world that looks like a cabin room with windows. They are sitting at a desk and can see their laptop screen as part of the virtual world.
  Interventions: Behavioral: Meta Quest 3 VR Headset with noise cancelling headphones
- Virtual Reality + Feedback (Experimental): Participants in this condition wear the virtual reality headset. They are emersed in a virtual world that looks like a cabin room with windows. They are sitting at a desk and can see their laptop screen as part of the virtual world. The program tracks their keyboard and mouse click data to assess how consistently they are working. A stoplight in the virtual environment is green when they are working consistently and turns red when the not.
  Interventions: Behavioral: Meta Quest 3 VR Headset with noise cancelling headphones

INTERVENTIONS:
Behavioral: Meta Quest 3 VR Headset with noise cancelling headphones — Wearing the headset and headphones removes all outside audio and visual distractions. One of the groups receives frequent and consistent feedback about work productivity similar to behavioral interventions for ADHD.

SUMMARY:
The goal of this pilot randomized clinical trial is to test the impact of a virtual reality program for improving the ability of emerging adults (age 18-25) with attention deficit hyperactivity disorder (ADHD) to stay focused while completing homework and studying. This study compares the impact of using a virtual reality headset to using a virtual reality headset while also receiving feedback about levels of focus to a control group. The main question is whether participants demonstrate significantly improved concentration while completing homework and studying in virtual reality and whether they enjoy and prefer working in a virtual reality environment. Concentration is measured both through participant report and also using keyboard and mouse click data to assess work productivity objectively.

DETAILED DESCRIPTION:
This study involves a pilot randomized control trial (RCT) to assess the feasibility/usability and preliminary effects of a virtual reality (VR) environment alone (n=15) compared to VR environment + feedback about focus (n=15) and to a VR passthrough control (n=15). Proposed mechanisms of action will be measured every session, including data on keyboard and mouse clicks plus self-ratings of concentration, homework effort, and homework motivation. After completing the initial diagnostic evaluation and confirming eligibility, 45 emerging adults with ADHD (ages 18-25) will be randomized to 1 of 3 groups and then provided with a VR headset and computer to use in their dorm/home. Randomization will be performed (1:1:1) to the three conditions. Randomization will be blocked on ADHD medication status to ensure an equal number of participants taking and not taking ADHD medication in each group. Phase 3 includes a 2-session baseline where all participants complete homework and study without using the VR headset.

Group 1, VR passthrough: After completing the two session baseline, participants will use the VR headset in their room/home or the library 10 times over two weeks (max twice a day with a minimum 2-hour break) for 1-hour sessions each time. The participant will wear the headset, but it will not be used as usual. The headset will be in "VR passthrough" mode, meaning the participant will see through to the normal environment and laptop (i.e., they can see the real world around them, just wearing a headset).

Group 2, VR environment only: After completing the two session baseline, participants will use the VR headset in their room/home or the library 10 times over two weeks (max twice a day with a minimum 2-hour break) for 1-hour sessions each time. For the following sessions, the participant will wear the VR headset and engage in homework in the VR environment.

Group 2, VR environment + feedback: After completing the two session baseline, participants will use the VR headset in their room/home or the 10 times over two weeks (max twice a day with a minimum 2-hour break) for 1-hour sessions each time. For the following sessions, the participant will wear the VR headset and engage in homework in the VR environment while receiving real time visual feedback on performance and focus.

Participants concentration, effort/efficiency, and motivation is assessed each baseline and VR session, and participants answer questions about VR feasibility, useability, and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* To be included, participants must meet DSM-5 criteria for ADHD and be between the ages of 18 and 25. Given high rates of comorbidities in college students with ADHD, participants who meet criteria for ODD, anxiety or depressive disorders on the diagnostic interview are not excluded. In addition, participants must have an item mean score of >2.0 (often or very often) on the homework task specific version of the Adult Concentration Index (ACI), ensuring the presence of a problem in the mechanism being targeted in this study. The participant has to endorse a total of at least 5 symptoms in the ADHD inattention domain as currently present and impairing and at least 6 symptoms in the ADHD inattention domain as present and impairing during childhood. To rule out exclusionary conditions and/or to assess for the presence of comorbid conditions, psychological functioning will be assessed using the DSM-5 version of the Structured Clinical Interview for DSM Disorders (SCID-5-RV)

Exclusion Criteria:

* Whether primary or not, the comorbid presence of several other conditions will be exclusionary. This includes autism spectrum disorders, bipolar disorder, obsessive-compulsive disorder, active substance abuse, and other psychiatric conditions whose treatment precludes participation in the study. Students who do not meet criteria for ADHD or who are not in the specified age range are also not eligible to participate. Students with a history of seizures are not eligible to participate given the use of VR.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Langberg, PhD, Principal Investigator — Rutgers University
Locations (2):
- United States (2):
  - Louisiana State University, Baton Rouge, Louisiana
  - Rutgers University - New Brunswick, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
De-identified data can be used for many secondary analyses. Individual subject-level data and item-level data will be shared. Prior to sharing, all data will be de-identified so that it is HIPAA-compliant. Once deposited into an open database, data will be open to the greater scientific community according to the terms of the individual database. Data will then be fully available for secondary analyses, data mining, and to facilitate discovery by combining our data with that of other centers/investigators for large-scale analyses. As we will be using the NDA, this repository has policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations. The NIMH Data Archive (NDA) will serve as the primary data repository for the current proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Analyzed/experimental data related to the primary aims of the study will be submitted when a publication on the data is accepted, or the project period ends, and shared when published or one year after the project period ends, whichever comes first in both cases.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We ask the participants their current ADHD medication status because we block randomize based on if they are taking medication or not, to ensure groups are well-balanced between taking medication and not taking medication.
Period: Overall Study
Arm/Group | VR Passthrough | Virtual Reality | Virtual Reality + Feedback
Started | 22 | 18 | 20
Completed (Milestone definition: Participants who made it to at least 7 sessions, which is milestone 1 out of 2.) | 16 | 16 | 17
Not Completed | 6 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VR Passthrough | Virtual Reality | Virtual Reality + Feedback | Total
Number analyzed (Participants) | 22 | 18 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants] — Participants were eligible if they were between the ages of 18-25
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 22 | 18 | 20 | 60
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 11 | 40
  Male | 7 | 4 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 6 | 10
  Not Hispanic or Latino | 20 | 16 | 14 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 6 | 13
  White | 15 | 11 | 12 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 18 | 20 | 60
The Barkley Adult Attention Deficit/Hyperactivity Disorder (ADHD) Rating Scale-IV Self-Report [Mean (Standard Deviation); unit: units on a scale] — Assesses ADHD symptoms in adults age 18+, aligning with symptoms that are used to diagnose ADHD in the DSM-5. Rating options;Never, Sometimes, Often, Very Often. Participants were given this survey via Redcap after viewing a recruitment flyer that had a QR code.Higher # = more severe ADHD symptoms. Total scores/symptom counts summed. Please see below for letters associated with subscales. Ranges of these subscales: A (0-9), B (0-27), C (0-9), D (0-27), E (0-27), F (0-81), G (0-9), H (0-27), I (0-9), J (0-27), K (0-18), L (0-54).
  units on a scale
    Current Inattention Symptom Count (A) | 7.27 (1.12) | 7.50 (1.58) | 7.15 (1.42) | 7.30 (1.36)
    Current Inattention Total Rating Score (B) | 19.59 (3.72) | 20.44 (3.67) | 19.80 (3.81) | 19.91 (3.69)
    Current Hyperactive Symptom Count (C) | 5.05 (1.96) | 4.94 (2.73) | 5.75 (1.55) | 5.25 (2.10)
    Current Hyperactive Total Rating Score (D) | 15.36 (4.28) | 15.89 (6.06) | 16.85 (3.51) | 16.02 (4.63)
    Current Total ADHD Symptom Count (E) | 18.32 (2.77) | 18.44 (5.14) | 18.35 (3.50) | 18.37 (3.78)
    Current Total ADHD Rating Score (F) | 52.09 (7.98) | 53.72 (11.90) | 52.60 (8.67) | 52.75 (9.39)
    Past Inattention Symptom Count (G) | 7.32 (2.19) | 7.33 (1.94) | 7.05 (1.64) | 7.23 (1.92)
    Past inattention Total Rating Score (H) | 19.91 (5.77) | 20.28 (4.55) | 19.95 (4.62) | 20.03 (4.97)
    Past hyperactive/impulsive Symptom Count (I) | 6.14 (2.29) | 5.17 (3.00) | 6.55 (1.82) | 5.98 (2.42)
    Past Hyper/Impulsive Total Rating Score (J) | 17.50 (5.69) | 15.78 (7.11) | 19.30 (4.40) | 17.58 (5.86)
    Past Total Adhd Symptom Count (K) | 13.45 (3.49) | 12.50 (4.44) | 13.60 (3.14) | 13.22 (3.66)
    Past Total ADHD Rating Score (L) | 37.41 (10.00) | 36.06 (10.71) | 39.25 (7.89) | 37.62 (9.50)
Adult Concentration Index (ACI) [Mean (Standard Deviation); unit: units on a scale] — Measures how true statements pertaining to concentration are. Includes "I can't focus, I daydream" as items.Distributed via redcap survey to ps eligible after completing BAARS. Rating options: Not at all, sometimes, often, very often.Totals include ACI symptom count range 0-7, ACI total rating score range 0-21.
  Higher # = more severe levels of difficulty concentrating. Sx ct scores and total rating scores are summed.
  units on a scale
    ACI Symptom Count | 5.91 (1.06) | 5.94 (1.30) | 6.35 (.81) | 6.07 (1.07)
    ACI Total Score | 16.05 (3.09) | 16.61 (3.76) | 17.65 (2.74) | 16.75 (3.22)
General Anxiety Disorder-7 (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — GAD-7 measures severity of anxiety in participants. Ps are given this survey via Redcap after they are eligible based on BAARS and ACI. There are no subscales in this instrument, only a total score. The rating options are Not at all, several days, more than half the days, nearly every day. Higher # = more severe levels of anxiety. Total score range 0-21. Scores are summed.
  units on a scale | 12.55 (3.31) | 10.11 (5.57) | 11.25 (4.89) | 11.38 (4.64)
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — This instrument measures depression and its severity. Participants received this survey if they were eligible based on the BAARS and ACI. There are no subscales in this measure, just a total score. The rating options are Not at all, several days, more than half the days, and nearly every day. Total score range 0-27. Higher values = worse depression symptom severity. Total scores are summed.
  units on a scale | 12.00 (6.90) | 9.83 (6.86) | 9.85 (5.08) | 10.63 (6.32)
Columbia Suicide Severity Rating Scale (C-SSRS) [Mean (Standard Deviation); unit: units on a scale] — The CSSRS is used for suicide risk assessment. Participants were given this survey via redcap if they were eligible based on the BAARS and ACI. The rating options are yes ( =1) /no (=0). There were no subscales for this measure, just a total score. The total score range is 0-6. Higher # = more risk for suicide. The total scores are summed. Population: The number of participants analyzed from the overall number is different because participants only complete the whole C-SSR if they answer 'yes' to question #2 - "Have you actually had any thoughts of killing yourself." If they answer yes, they are brought to 4 more questions which is totaled for the score reported. Those 4 other questions are about actual suicide attempts, which we wouldn't ask about if a participant did not think about suicide in the first place.
  units on a scale
    number analyzed (Participants) | 7 | 4 | 3 | 14
    (all) | 3.14 (1.77) | 3.25 (1.26) | 4.0 (1.00) | 3.36 (1.45)
Barkley Deficits in Executive Functioning Scale (BDEFS-Short Form) [Mean (Standard Deviation); unit: units on a scale] — BDEFS measures executive functioning in adults. Participants were given this survey via Redcap if they were eligible based on the BAARS and ACI. The rating options are Never or Rarely, Sometimes, Often, and Very Often. There are no subscales for this measure, only totals. They are BDEFS symptom count - range 0-20, and BDEFS total rating score - range 20-80. Higher #s = worse executive functioning outcome. Total scores are summed.
  units on a scale
    BDEFs Symptom Count | 17.55 (2.69) | 17.28 (3.01) | 17.35 (2.37) | 17.40 (2.64)
    BDEFs Total Rating Score | 53.82 (7.63) | 55.67 (13.50) | 56.3 (11.15) | 55.20 (10.70)
Barkley Functional Impairment Scale (BFIS) [Mean (Standard Deviation); unit: scores on a scale] — BFIS measures possible impairment in 15 major domains of psychosocial functioning in adults. Participants were given this survey via redcap if they were eligible based on the BAARS and ACI. There are no subscales in this measure. Answer choices are on a scale: 0 = Not at All, 1-2 = Somewhat, 3-4 =Mild, 5-7 = Moderate, 8-9 = Severe. The total score is a mean with a range of 0-9. Higher #s = worse domains of functioning.
  scores on a scale | 4.91 (1.52) | 4.62 (1.75) | 4.42 (2.00) | 4.66 (1.74)
Baseline Homework Motivation Index [Mean (Standard Deviation); unit: units on a scale] — This measure of motivation level for completing homework has rating options which include Not True, Somewhat True, Pretty Much True, and Definitely True. Participants were given this survey via Redcap if they were eligible based on the BAARS and ACI. There are no subscales, just a total measure. Range is 7-28. Higher # = better motivation levels to complete homework. Total scores are summed.
  units on a scale | 19.55 (4.24) | 20.17 (4.49) | 19.85 (3.22) | 19.83 (3.95)
Baseline Homework Effort Index [Mean (Standard Deviation); unit: units on a scale] — This measure looks at how much effort participants put into their homework. The rating options are Not True, Somewhat True, Pretty Much True, and Definitely True. Participants were given this survey via Redcap if they were eligible based on the BAARS and ACI. There are no subscales in this measure, just a total score. The range is 7-28. Higher #s = better effort levels to complete homework. The total score is summed.
  units on a scale | 17.09 (3.83) | 16.50 (4.62) | 15.80 (4.53) | 16.48 (4.27)

OUTCOME MEASURES:

1. Primary Outcome: Objective On-Task Assessment Algorithm
Description: Percentage of time on-task during each study session utilizing the Objective On-Task Assessment algorithmic mouse and keyboard click data.
  There are no subscales in this measure. Percentages below are for sessions 1-2 (T1) and 3-12 (T2). Participants had 2 weeks to complete sessions 1-7 and a 3rd week to complete the last 5 sessions (sessions 8-12), equaling 12 sessions within 3 weeks. The 1-7 and 8-12 time points were only for compensation/motivational purposes (payment after sessions 1-7 and after 8-12) and were not outcome measurement time points. Sessions 1+2 are combined for a time point because participants did not wear headsets for those two sessions, which we considered 'baseline,' giving us a base focus score before participants put on a headset. Participants wore the headsets for sessions 3-12. Percentages below were averaged for each time point. T1 is an average of session 1+2's percentages. T2 is an average of sessions 3-12's percentages.
Time Frame: Participants had 2 weeks to complete sessions 1-7 and a 3rd week to complete the last 5 sessions, equaling 12 sessions within 3 weeks.
Population: Number of participants analyzed differs between the overall number analyzed as some participants did not complete enough sessions or the sessions were faulty, and they were excluded from this measure. The number analyzed here is even less than the other outcome measures as it is easier to get measure information through surveys if a session is faulty, over the whole focus algorithm, which doesn't capture information if there are glitches in the virtual reality system.
Measure: Mean (Standard Deviation); unit: percentage of time focused
Arm/Group | VR Passthrough | Virtual Reality | Virtual Reality + Feedback
Number analyzed (Participants) | 22 | 18 | 20
percentage of time focused
  Sessions 1+2 (T1)(Baseline): number analyzed (Participants) | 16 | 14 | 14
  Sessions 1+2 (T1)(Baseline) | .86 (.21) | .62 (.35) | .83 (.27)
  Sessions 3-12 (T2): number analyzed (Participants) | 16 | 14 | 14
  Sessions 3-12 (T2) | .83 (.04) | .85 (.06) | .95 (.01)

2. Primary Outcome: Homework Concentration Index
Description: This measure looks at how concentrated participants were while completing their homework.The rating options are Not True, Somewhat True, Pretty Much True, and Definitely True. There are no subscales in this measure, just a total score. The range is 7-28. Higher #s = worse concentration. The total score is summed. Numbers below are averages of units from sessions 1-2 (T1) and 3-12 (T2).The units were collected during each session's post survey. Sessions 1+2 are combined for a time point because participants did not wear headsets for those two sessions. Participants wore the headsets for sessions 3-12. Sessions 1+2 are considered baseline as they gave us a baseline score before participants put on a headset. Scores below were averaged for T1 (Sessions 1+2) and T2 (Sessions 3-12).
Time Frame: Participants had 2 weeks to complete sessions 1-7, a 3rd week to complete the last 5 sessions (sessions 8-12), equaling 12 sessions within 3 weeks.The 1-7 and 8-12 time points were only for compensation purposes and were not outcome measure points.
Population: Number of participants analyzed differs between timepoints as some participants did not complete enough sessions or the sessions were faulty, and they were excluded from T2. Some participants also dropped out after 2 sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VR Passthrough | Virtual Reality | Virtual Reality + Feedback
Number analyzed (Participants) | 22 | 18 | 20
units on a scale
  Sessions 1+2 (T1)(Baseline) | 15.93 (4.69) | 16.17 (6.03) | 17.93 (5.57)
  Sessions 3-12 (T2): number analyzed (Participants) | 20 | 18 | 19
  Sessions 3-12 (T2) | 11.82 (5.19) | 12.75 (3.88) | 12.96 (4.37)

3. Secondary Outcome: Homework Effort Index
Description: The Homework Effort Index looks at how much effort participants were able to put in while completing their homework.The rating options are Not True, Somewhat True, Pretty Much True, and Definitely True. There are no subscales in this measure, just a total score. The range is 7-28. Higher #s = greater levels of effort. The total score is summed. Scores below are averages of units from sessions 1-2 (T1) and 3-12 (T2).The units were collected during each session's post survey. Sessions 1+2 are combined for a time point because participants did not wear headsets for those two sessions. Participants wore the headsets for sessions 3-12. Sessions 1+2 are considered baseline as they gave us a baseline score before participants put on a headset. Scores below are averaged for T1 and T2.
Time Frame: Participants had 2 weeks to complete sessions 1-7, a 3rd week to complete the last 5 sessions (sessions 8-12), equaling 12 sessions within 3 weeks. The 1-7 and 8-12 time points were only for compensation purposes and were not outcome measure points.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VR Passthrough | Virtual Reality | Virtual Reality + Feedback
Number analyzed (Participants) | 22 | 18 | 20
units on a scale
  Sessions 1+2 (T1)(Baseline) | 19.34 (3.93) | 17.69 (3.06) | 17.43 (3.05)
  Sessions 3-12 (T2): number analyzed (Participants) | 19 | 18 | 19
  Sessions 3-12 (T2) | 19.95 (5.31) | 19.63 (4.42) | 19.92 (5.08)

4. Secondary Outcome: Homework Motivation Index
Description: The Homework Motivation Index measures how motivated participants were while completing their homework.The rating options are Not True, Somewhat True, Pretty Much True, and Definitely True.There are no subscales in this measure, just a total score. The range is 7-28. Higher #s = greater levels of motivation. The total score is summed.
  Scores below are averages of units from sessions 1-2 (T1) and 3-12 (T2).The units were collected during each session's post survey. Sessions 1+2 are combined for a time point because participants did not wear headsets for those two sessions. Participants wore the headsets for sessions 3-12. Sessions 1+2 are considered baseline as they gave us a baseline score before participants put on a headset. Scores below were averaged for T1 and T2.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VR Passthrough | Virtual Reality | Virtual Reality + Feedback
Number analyzed (Participants) | 22 | 18 | 20
units on a scale
  Sessions 1+2 (T1)(Baseline) | 20.73 (4.20) | 19.94 (3.40) | 19.35 (3.21)
  Sessions 3-12 (T2): number analyzed (Participants) | 20 | 18 | 19
  Sessions 3-12 (T2) | 21.08 (6.89) | 20.53 (5.30) | 20.89 (5.07)

ADVERSE EVENTS:
Time Frame: AE data was monitored over 1-2 months, including the baseline assessment and active phase of the study with the VR sessions. Whether it was 1 or 2 months depended on how long participants took to schedule their baseline assessment, to pick up their VR technology, to complete the 12 sessions.We were in regular contact with participants over the time frame to ask how they were adjusting to the VR and to see if they had any problems.No participants met the criteria for adverse events in our study.
Description: During the preliminary baseline surveys which were administered before the assessment, there is a questionnaire asking about a participant's medical history. If participants answered yes to this question: "Do you have any conditions where flashing or intense light might affect you, such as epilepsy, migraines, unexplained seizures, recent concussions, or light sensitivity," they were not eligible to continue with the study. This exclusion was agreed upon with our IRB.
Arm/Group | VR Passthrough | Virtual Reality | Virtual Reality + Feedback
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT06454604/Prot_SAP_001.pdf
  • Informed Consent Form (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT06454604/ICF_002.pdf